CLINICAL TRIAL: NCT00570856
Title: Clinical Trial of Effectiveness of Folic Acid Therapy on Homocysteine Level and Carotid Intima-Media Thickness After Kidney Transplantation
Brief Title: Trial of Folic Acid Effect on Hcy and cIMT After Kidney Tx
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Dr. Mohsen Nafar, Shaheed Beheshti Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 110; 110
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-12

CONDITIONS: Kidney Transplantation
Keywords: Folic Acid; Homocysteine; intima-media thickness
MeSH Terms: interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Folic acid supplementation
  Interventions: Drug: Folic acid
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Folic acid — Folic acid 5 mg/day
  Arms: 1
Drug: Placebo — Placebo similar to the folic acid tablets, 1/day
  Arms: 2

SUMMARY:
To see the effect of Folic acid supplementation after kidney transplantation on plasma total homocysteine level and carotid intimal-media thickness

ELIGIBILITY:
Inclusion Criteria:

* having hyperhomocysteinemia(tHcy>12.5 µmol/L in men and 11.5 µmol/L in women )
* No evident history of CVD 4. no evidence of cigarette smoking
* not participating in other clinical studies on evaluation of cardiac diseases and
* not taking any lipid lowering treatment
* not being pregnant or breast feeding a baby(women)
* Having HIV or viral hepatitis infections.

Exclusion Criteria:

* unstable condition of the transplanted kidney (Cr> 3 mg/dl, BUN > 50 mg/dl)
* Cyclosporine (CsA) intoxication
* New onset of any severe disease ( such as MI, stroke, DM, etc.).

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-06; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
plasma level of total homocysteine (tHcy) | 6 months

SECONDARY OUTCOMES:
carotid intima-media thickness (cIMT) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Nafar, MD- Nephrologist, Study Chair — Urology Nephrology Research Center, Labbafi Nejad Hospital, Shaheed Beheshti University of Medical Sciences, Tehran, Iran; Farideh Khatami, Master of Science, Principal Investigator — Labbafi Nejad Hospital, Shaheed Beheshti University of Medical Sciences, Tehran, Iran; Babak Kardavani, M.D., Principal Investigator — Urology Nephrology Research Center, Labbafi Nejad Hospital, Shaheed Beheshti University of Medical Sciences, Tehran, Iran